CLINICAL TRIAL: NCT05787509
Title: The Exploration of Prolonged Treatment With Vaginal Progesterone to Prevent Preterm Birth From IVF Fresh Embryo Transplantation Cycle: a Randomized Controlled Trial
Brief Title: Prolonged Progesterone to Prevent Preterm Birth From IVF - ET
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSKY-2022-389-01
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Trial group (Experimental): we will prolong the duration of vaginal progesterone treatment until 24 weeks of gestation.
  Interventions: Drug: Progesterone Sustained-release vaginal gel
- The control group (Experimental): we will use vaginal progesterone treatment until 12 weeks of gestation.
  Interventions: Drug: Progesterone Sustained-release vaginal gel

INTERVENTIONS:
Drug: Progesterone Sustained-release vaginal gel — the treatment time of vaginal progesterone
  Other Names: Vaginal progesterone

SUMMARY:
To investigate the incidence of preterm birth in IVF fresh embryo transplantation cycle patients after prolonged vaginal progesterone treatment

DETAILED DESCRIPTION:
Participant: 20-40 years old, IVF fresh embryo transplantation, singleton pregnancy, blood/urine HCG (+) Control group: The administration of vaginal progesterone (90mg/d) began from positive HCG in blood/urine until 12 weeks of gestation. Regular delivery examinations were conducted, and cervical length was detected by B-ultrasound at 12, 16, 20 and 24 weeks of gestation respectively, while fetal growth and development were monitored. Follow-up was continued until the end of delivery.

Trial group: The administration of vaginal progesterone (90mg/d) began from positive HCG in blood/urine until 24 weeks of gestation. Regular delivery examinations were conducted, and cervical length was detected by B-ultrasound at 12, 16, 20 and 24 weeks of gestation respectively, while fetal growth and development were monitored. Follow-up was continued until the end of delivery.

Observation index: The gestational age of delivery, symptoms of preterm birth and gestational age, gestational age at preterm birth or abortion, fetal growth and development, neonatal outcomes, and drug-related adverse reactions were recorded for each participant.

ELIGIBILITY:
Inclusion Criteria:

* 1. 20-40 years old 2. met the conditions of assisted reproductive technology and underwent IVF fresh embryo transplantation 3. Singleton pregnancy 4. Patients volunteered and signed informed consent prior to the trial.

Exclusion Criteria:

* 1. >40 years old 2. History of miscarriage or cervical insufficiency in the second trimester 3. Abnormal ovarian function or surgical history: decline in ovarian reserve, premature ovarian failure, Turner's syndrome, ovarian cyst excision, PCOS perforation/coning, chocolate cyst surgery, ovarian cone resection 4. Uterine deformities: including single horn uterus, double horn uterus, residual horn uterus, saddle uterus, infantile uterus, double uterus, mediastinal uterus 5. Diseases affecting uterine shape: uterine adhesions, uterine submucosal myomas or polyps, adenomyosis, chronic inflammation of the endometrium 6. Abnormalities in cervical morphology or function. 7. History of total cervicectomy, conical excision, and cervical insufficiency 8. Vaginal inflammation: refractory candida vaginitis, bacterial vaginosis, persistent mycoplasma-positive vaginosis, persistent chlamydia-positive vaginosis 9. B ultrasonography indicates twin or multiple pregnancies 10. Patients with severe medical and surgical diseases 11. Participants who had participated in other clinical trials during the 90 days or had received any investigational clinical drug during the 30 days prior to the trial 12. Patients with no long-term follow-up or poor compliance 13. The investigator believes that there are any factors that may affect participants' participation in the study or the evaluation of the results

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of preterm birth | 37 weeks of gestation
  the symptom or diagnosis of preterm birth

IPD SHARING:
Plan to Share IPD: No